CLINICAL TRIAL: NCT03044912
Title: Therapeutic Efficacy and Safety of Mirabegron , a β3-Adrenoceptor Agonist, Treatment on Patients With Overactive Bladder Syndrome in Taiwan - Comparison of Therapeutic Efficacy and Safety Between 25mg and 50mg
Brief Title: Therapeutic Efficacy and Safety of Mirabegron Treatment on Patients With Overactive Bladder Syndrome in Taiwan
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Buddhist Tzu Chi General Hospital (Other)
Responsible Party: Principal Investigator, Hann-Chorng Kuo, Chairman and Professor, Department of Urology, Buddhist Tzu Chi General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TCGHUROL012
Record Dates: First submitted 2017-02-03; First posted 2017-02-07 (Estimated); Last update posted 2017-02-09 (Estimated); Status verified 2017-02

CONDITIONS: Overactive Bladder Syndrome
MeSH Terms: interventions — mirabegron

STUDY DESIGN:
Intervention Model Description: Randomized open label study
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- treatment group (Experimental): Mirabegron 50 mg for comparison
  Interventions: Drug: mirabegron
- Comparative group (Active Comparator): Patient take Mirabegron 25 mg
  Interventions: Drug: mirabegron

INTERVENTIONS:
Drug: mirabegron — To evaluate the efficacy and safety of Mirabegron 50 mg vs 25 mg in Taiwanese patients with overactive bladder syndrome
  Other Names: Betmiga

SUMMARY:
Recent phase III trials have confirmed the efficacy and safety of mirabegron in the treatment of overactive bladder (OAB) in Europeans, Australians, North Americans, Japanese and Asians. Whether mirabegron 25mg or 50mg should be used as the first line treatment for OAB has not been determined yet. The dose effectiveness relationship between 25mg and 50mg mirabegron has also not been investigated yet. Hence, investigators have conducted this post marketing study in order to evaluate the efficacy and safety between mirabegron 25mg and 50mg in Taiwanese people with symptoms of OAB.

DETAILED DESCRIPTION:
Overactive bladder syndrome (OAB) is defined as the symptom syndrome with frequency, and urgency with or without urgency incontinence. OAB affects more than 400 million people worldwide and has been estimated to affect around 16% of the adult population across Europe and the USA. In Asian countries, the prevalence of OAB has been reported to be 6% of men and women aged ≥18 years in China; 12.2% of men and women in Korea;12.4% of men and women aged ≥40 years in Japan; and 21 to 25% of women and 16.9% of community dwelling adults in Taiwan. Another study reported that the prevalence of OAB among adult men across 11 Asian countries (India, Indonesia, Malaysia, Pakistan, Philippines, Singapore, South Korea, Taiwan, China, Hong Kong and Thailand) was 29.9%.

Antimuscarinics are first line pharmacotherapy for OAB. However, some patients have a suboptimal response to antimuscarinics and some may experience adverse effects, such as dry mouth or constipation. Therefore, a high proportion of patients discontinue antimuscarinic therapy, with fewer than 25% remaining on treatment at 1 year. There is an unmet need to develop new drugs for OAB without the bothersome adverse effects of antimuscarinic agents.

β3-adrenergic receptors are known to promote urine storage in the bladder by inducing detrusor relaxation in animal and human bladders. In humans, the β3-adrenoceptor is the predominant β-receptor subtype in the urinary bladder. β3-adrenoceptor agonists relax the detrusor smooth muscle during the bladder storage phase and increase bladder capacity without accompanying changes in micturition pressure, residual volume or voiding contraction.

Mirabegron is the first β3-adrenoceptor agonist to have been approved for the treatment of OAB. Pooled safety data indicates that dry mouth, the chief cause of treatment discontinuation with antimuscarinic agents, occurs with low incidence with mirabegronc. Hence, mirabegron may be a valuable treatment option for patients with OAB.

Recent phase III trials have confirmed the efficacy and safety of mirabegron in the treatment of OAB in Europeans, Australians, North Americans, Japanese and Asians. Whether mirabegron 25mg or 50mg should be used as the first line treatment for OAB has not been determined yet. The dose effectiveness relationship between 25mg and 50mg mirabegron has also not been investigated yet. Hence, investigators have conducted this post-marketing study in order to evaluate the efficacy and safety between mirabegron 25mg and 50mg in Taiwanese people with symptoms of OAB.

Materials and Methods

Study Title: Therapeutic Efficacy and Safety of Mirabegron , a β3-Adrenoceptor Agonist, for Patients with Overactive Bladder Syndrome in Taiwan

Primary objective: to evaluate the efficacy of Mirabegron 50 mg vs 25 mg in Taiwanese patients

Secondary objective: to assess safety and tolerability of Mirabegron 50 mg vs 25 mg in Taiwanese patients

Other objective: to investigate potential predictive factors of treatment outcome using baseline demographic (ex. Comorbidity, age, etc.) and urodynamic study findings.

Randomization will be accomplished using a computer-generated randomization scheme (Cenduit GmbH, Allshwil, Switzerland) with stratification by site; allocation to treatment groups at each site was accomplished via an interactive response system with a study coordinator. Study visits took place at Week 0 (Visit 1; confirmation of eligibility criteria); Weeks 4, 8 and 12 (Visits 2, 3 and 4).

The study will be approved by the institutional review board of each study site and conducted in accordance with the ethical principles that have their origin in the Declaration of Helsinki, Good Clinical Practice, International Conference on Harmonisation guidelines, and all applicable laws and regulations.

Efficacy End-points:

Primary endpoint(s): The percentage of patients with a change from baseline to the final visit in the urgency episodes per 24 hours by 2 or greater.

Secondary endpoint(s):

1. Secondary efficacy end-points are change from baseline to the final visit in OABSS score, Patient Perception on Intensity of Urgency Scale (PPIUS), mean number of frequency episodes, urinary incontinence episodes, urgency incontinence episodes and nocturia episodes per 24 hours, and mean volume voided per micturition. Change from baseline to each study visit in each efficacy variable will also be measured. An additional secondary end-point is change from baseline to final visit in the Patient Perception of the ladder Condition (PPBC) to assess patients' subjective satisfaction of treatment drugs on bladder conditions. Paper diary will be used in this trial.
2. Adverse events (AEs) are assessed at all visits. Safety endpoints are incidence and severity of AEs, and changes from baseline to end-of-treatment in vital signs (heart rate, systolic and diastolic blood pressures) and laboratory tests (hematology, biochemistry and urinalysis).
3. To determine the predictive factors of treatment outcome using baseline demographic (ex. comorbidity, age, etc.) and urodynamic study findings.

PPIUS (Patient Perception of Intensity of Urgency Scale):

0. No urgency, I felt no need to empty my bladder, but did so for other reasons.

1. Mild urgency, I could postpone voiding as long as necessary, without fear of wetting myself.
2. Moderate urgency, I could postpone voiding for a short while, without fear of wetting myself.
3. Severe urgency, I could postpone voiding, but had to rush to the toilet in order not to wet myself.
4. Urge incontinence, I leaked before reaching the toilet.

Patient Perception of the ladder Condition (PPBC):

Which of the following statements describes your bladder condition best at the moment? 0: My bladder condition does not cause me any problems at all.

1. My bladder condition causes me some very minor problems.
2. My bladder condition causes me some minor problems.
3. My bladder condition causes me (some) moderate problems.
4. My bladder condition causes me severe problems.
5. My bladder condition causes me many severe problems.

Safety Assessment:

Safety assessments included reporting of adverse events (AEs, all unfavorable signs and symptoms observed from the start of the run-in period until the end of the follow-up period). Exacerbation of the symptoms of OAB was not defined as an AE in this clinical study.

Sample size: 574 patients within two years Justification:The sample size for this study was based on results from a 12-week Phase III study (178-CL-074). In 074 study, the responder analysis for reduction in urgency episodes for minimum important difference of 1.54 episodes was 47.1% in the M25 group and 57.7% in the M50 group. In this ISR, the primary efficacy end-point is the percentage of patients with a change from baseline to the final visit in the urgency episodes per 24 hours by 2 or greater. The responding rate is assumed as 60% in the M50 group and 45% in the M25 group. The number of patients per group necessary to demonstrate superiority to the first group (mirabegron 25mg for 12 weeks) would be 244 at a two-sided significance level of 5% and power of 90%. Assuming a dropout rate of 15% during the treatment period, 287 subjects per group are to be enrolled for randomization.

Expected Results:

The results of this study will demonstrate that:

1. Mirabegron 25mg once-daily for 12 weeks is effective and safe in treatment of patients with OAB (group 1).
2. Mirabegron 50mg is effective in improving OAB symptoms when the therapeutic efficacy of the dose of 25mg mirabegron for 4 weeks is suboptimal (group 2)
3. Investigators will try to search for predictive factors for responders to mirabegron 25mg alone, escalating to mirabegron 50mg, based on the baseline demographics and urodynamic study findings,

ELIGIBILITY:
Inclusion Criteria:

1. symptoms of OAB for at least 12 weeks before initiation of the run-in period;
2. an average of ≥8 micturitions per 24 hours,
3. an average of ≥2 episode of urgency or urgency incontinence per 24-hours, during a 3-day micturition diary period.
4. no prior pharmacological treatment for OAB

Exclusion Criteria:

1. stress urinary incontinence as a predominant symptom at screening;
2. urinary tract infection, urinary stone, interstitial cystitis or a history of recurrent urinary tract infection;
3. confirmed post-void residual (PVR) volume of ≥100 mL or more or with a clinically significant lower urinary tract obstructive disease;
4. proven neurogenic bladder such as spinal cord injury, multiple sclerosis;
5. overt bladder outlet obstruction.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 574 (Estimated)
Dates: Start 2015-11-16 (Actual); Primary Completion 2019-02-01 (Estimated); Study Completion 2019-08-01 (Estimated)

PRIMARY OUTCOMES:
Changes of urgency episodes by 2 per 24 hours | baseline and 3 months
  The percentage of patients with a change from baseline to the final visit in the urgency episodes per 24 hours by 2 or greater

SECONDARY OUTCOMES:
Net change of overactive bladder symptom score (OABSS) | baseline and 3 months
  Net change from baseline to the final visit in OABSS score
Patient Perception on Intensity of Urgency Scale (PPIUS) | baseline and 3 months
  Net change of Patient Perception on Intensity of Urgency Scale (PPIUS) from baseline to the final visit
Net change of mean number of frequency episodes | baseline and 3 months
  The net change of mean number of frequency episodes from baselinbe to the final visit
The net change of mean number of urinary incontinence episodes | baseline and 3 months
  The net change of mean number of urinary incontinence episodes from baseline to the final visit
Net change of the mean number of urgency incontinence episodes | baseline and 3 months
  Net change of the mean number of urgency incontinence episodes from baseline to the final visit
The net change of mean number of nocturia episodes per 24 hours | baseline and 3 months
  The net change of mean number of nocturia episodes per 24 hours from baselinev to the final visit
The net change of mean volume voided per micturition | baseline and 3 months
  The net change of mean volume voided per micturition from baseline to the final visit
The net change of the Patient Perception of the Bladder Condition (PPBC) | baseline and 3 months
  The net change in the Patient Perception of the Bladder Condition (PPBC) from baseline to final visit

CONTACTS AND LOCATIONS:
Overall Officials: Hann-Chorng Kuo, M.D., Study Director — Buddhist Tzu Chi General Hospital, Hualien, Taiwan
Locations (1):
- Buddhist Tzu Chi General Hospital, Hualien City, Taiwan

IPD SHARING:
Plan to Share IPD: No
IPD is not planned to be available